CLINICAL TRIAL: NCT00518687
Title: A Randomized, Multicenter, Double-Blind, Group-Sequential Study to Evaluate the Efficacy, Immunogenicity, and Safety of a Single Dose of Merck 0657nI Staphylococcus Aureus Vaccine (V710) in Adult Patients Scheduled for Cardiothoracic Surgery
Brief Title: Efficacy, Immunogenicity, and Safety of a Single Dose of V710 in Adult Patients Scheduled for Cardiothoracic Surgery (V710-003 AM2)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V710-003; 2007_523 (Other: Merck)
Record Dates: First submitted 2007-08-17; First posted 2007-08-21 (Estimated); Results first posted 2012-11-05 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Staphylococcus Aureus; Bacteremia; Mediastinitis
MeSH Terms: conditions — Staphylococcal Infections; Bacteremia; Mediastinitis | interventions — V710 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- V710 60 µg (Experimental)
  Interventions: Biological: V710
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: V710 — 0.5-mL single injection of V710 (60 µg)
  Other Names: Merck 0657nI Staphylococcus aureus vaccine
  Arms: V710 60 µg
Biological: Placebo — 0.5-mL single injection of matching placebo
  Arms: Placebo

SUMMARY:
This study will assess the efficacy of a single dose of V710 vaccine to prevent serious Staphylococcus aureus infections following elective cardiothoracic surgery. The study will also evaluate the immune response and general safety of the V710 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Participant is scheduled to undergo cardiothoracic surgery involving a full median sternotomy (not including cardiac transplantation surgery) within 14 to 60 days after vaccination.
* Female participants of reproductive potential are required to have a negative urine or serum pregnancy test immediately prior to study vaccination and must use an acceptable form of birth control.

Exclusion Criteria:

* Participants had an invasive Staphylococcus aureus infection within the past 3 months prior to study entry.
* A realistic (>50%) possibility that cardiothoracic surgery will be necessary sooner than 10 days after vaccination.
* Participant is planning to undergo cardiac transplantation surgery or sternal debridement to remedy an infection resulting from a prior cardiothoracic surgery.
* Participant has any type of ventricular-assist device in place at the time of study entry.
* Participant has a history of anaphylaxis to any of the vaccine components.
* Participant received V710 vaccine, any other investigational Staphylococcus aureus vaccine, or investigational Staphylococcus aureus antibodies.
* Participant has a temperature of ≥100.4ºF (≥38.0ºC), oral equivalent, within 48 hours prior to study vaccination.
* Participant has impairment of the immune system.
* Participant has a medical condition in which the expected survival is less than 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8031 (Actual)
Dates: Start 2007-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

REFERENCES:
- [Derived] Fowler VG, Allen KB, Moreira ED, Moustafa M, Isgro F, Boucher HW, Corey GR, Carmeli Y, Betts R, Hartzel JS, Chan IS, McNeely TB, Kartsonis NA, Guris D, Onorato MT, Smugar SS, DiNubile MJ, Sobanjo-ter Meulen A. Effect of an investigational vaccine for preventing Staphylococcus aureus infections after cardiothoracic surgery: a randomized trial. JAMA. 2013 Apr 3;309(13):1368-78. doi: 10.1001/jama.2013.3010. PMID 23549582

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo : 0.5-ml single injection of matching placebo
Period: Overall Study
Arm/Group | V710 60 µg | Placebo
Started | 4005 (An additional 10 participants were not analyzed because of questionable clinical practices at 1 site) | 4005 (An additional 11 participants were not analyzed because of questionable clinical practices at 1 site)
Vaccinated | 3981 | 3982
Completed | 2568 | 2585
Not Completed | 1437 | 1420
Not completed — Adverse Event | 201 | 177
Not completed — Lost to Follow-up | 144 | 155
Not completed — Physician Decision | 42 | 48
Not completed — Progressive disease | 2 | 2
Not completed — Protocol Violation | 8 | 10
Not completed — Study terminated by sponsor | 930 | 918
Not completed — Withdrawal by Subject | 110 | 110

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V710 60 µg | Placebo | Total
Number analyzed (Participants) | 4005 | 4005 | 8010
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (12.6) | 63.9 (12.5) | 63.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1328 | 1336 | 2664
  Male | 2677 | 2669 | 5346

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Staphylococcus Aureus Bacteremia and/or Deep Sternal Wound Infection
Description: Diagnosis of the Staphylococcus aureus infections employed standardized definitions adapted from the Centers for Disease Control (CDC) Guidelines for Nosocomial infections (Garner JS, Jarvis WS, Emori TG, et al. CDC definitions for nosocomial infections. APIC Infect Control App Epidemiol 1996;A1-20). Bacteremia was defined as ≥1 positive blood culture for S. aureus regardless of the presence of clinical symptoms. A Staphylococcus aureus deep sternal wound infection included mediastinitis or a deep incisional surgical-site infection involving the sternal wound.
Time Frame: Up to 90 days after surgery
Population: The population analyzed was the full analysis set: participants who were vaccinated and subsequently underwent cardiothoracic surgery involving full median sternotomy at least 14 days and at most 60 days after vaccination
Measure: Number; unit: participants
Arm/Group | V710 60 µg | Placebo
Number analyzed (Participants) | 3528 | 3517
participants | 22 | 27
Statistical Analysis 1: Comparison: V710 60 µg vs Placebo; Test type: Superiority or Other; p = 0.584, Exact 1-sided binomial test — A 1-sided p-value <0.025 implies that the V710 vaccine efficacy is statistically significantly greater than 20%; Vaccine Efficacy (VE) = 18.5, 95% CI 2-sided [-48.6 to 55.8] — VE = 1 - Relative Risk of V710 compared with placebo

2. Primary Outcome: Incidence Rate of Vaccine-related Serious Adverse Experiences
Description: Vaccine-related adverse experiences were those deemed by the investigator to be possibly, probably, or definitely vaccine related. A serious adverse experience was any adverse experience occurring at any dose that 1) resulted in death, 2) was life threatening, 3) resulted in a persistent or significant disability/incapacity, 4) resulted in or prolonged an existing inpatient hospitalization, 5) was a congenital anomaly/birth defect, 6) was a cancer, 7) was an overdose, or 8) jeopardized the participant and required medical or surgical intervention.
Time Frame: Up to 360 days after surgery
Population: The population analyzed included all vaccinated participants with follow-up results
Measure: Number; unit: Events per 100 person-years
Arm/Group | V710 60 µg | Placebo
Number analyzed (Participants) | 3958 | 3967
Events per 100 person-years | 0.0 | 0.0
Statistical Analysis 1: Comparison: V710 60 µg vs Placebo; Test type: Superiority or Other; p = 0.997, Miettinen and Nurminen; Estimated rate difference = 0.0, 95% CI 2-sided [-0.1 to 0.1]

3. Secondary Outcome: Number of Participants With Invasive Staphylococcus Aureus Infection
Description: Diagnosis of the Staphylococcus aureus infections employed standardized definitions adapted from the CDC Guidelines for Nosocomial infections. An invasive Staphylococcus infection included bacteremia, deep sternal wound infection, deep-tissue organ/space infection at another surgical site, or any other deep-tissue infection.
Time Frame: Up to 90 days after surgery
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | V710 60 µg | Placebo
Number analyzed (Participants) | 3528 | 3517
participants | 27 | 31
Statistical Analysis 1: Comparison: V710 60 µg vs Placebo; Test type: Superiority or Other; p = 0.347, Exact 1-sided binomial test — A 1-sided p-value <0.025 implies that the V710 vaccine efficacy is statistically significant; Vaccine Efficacy (VE) = 12.9, 95% CI 2-sided [-50.8 to 50.0] — VE = 1 - Relative Risk of V710 compared with placebo

4. Secondary Outcome: Number of Participants With Surgical-site Staphylococcus Aureus Infection
Description: Diagnosis of the Staphylococcus aureus infections employed standardized definitions adapted from the CDC Guidelines for Nosocomial infections. A Staphylococcus infection surgical-site infection included any superficial incisional, deep incisional, or organ/space infection at the sternal site, the vascular harvest (donor) site, or any other site at which the surgery was performed.
Time Frame: Up to 90 days after surgery
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | V710 60 µg | Placebo
Number analyzed (Participants) | 3528 | 3517
participants | 53 | 75
Statistical Analysis 1: Comparison: V710 60 µg vs Placebo; Test type: Superiority or Other; p = 0.032, Exact 1-sided binomial test — A 1-sided p-value <0.025 implies that the V710 vaccine efficacy is statistically significant; Vaccine Efficacy (VE) = 29.3, 95% CI 2-sided [-1.8 to 51.2] — VE = 1 - Relative Risk of V710 compared with placebo

ADVERSE EVENTS:
Time Frame: All serious adverse events (SAEs): through Day 14 after vaccination; vaccine-related SAEs, SAEs resulting in death, and SAEs involving infection diagnosis: through Day 360 after surgery; other adverse events (AEs): through Day 14 after vaccination
Description: The population analyzed was all vaccinated participants with follow-up results
Groups:
- V710 (60 µg) Lyophilized: V710: 0.5-ml single injection of V710 (60 µg)
Arm/Group | V710 (60 µg) Lyophilized | Placebo
Serious Adverse Events (participants affected / at risk) | 291/3958 | 274/3967
Other Adverse Events (participants affected / at risk) | 749/3958 | 343/3967
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V710 (60 µg) Lyophilized (N=3958) | Placebo (N=3967)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 6 (6) | 11 (11)
Angina pectoris (Cardiac disorders) | 3 (3) | 1 (1)
Angina unstable (Cardiac disorders) | 4 (4) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 18 (18) | 21 (21)
Cardiac failure (Cardiac disorders) | 12 (12) | 6 (6)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 5 (5) | 5 (5)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac ventricular disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 8 (8) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 23 (23) | 18 (18)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Low cardiac output syndrome (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3) | 8 (8)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 2 (2) | 5 (5)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1)
Ventricle rupture (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular dysfunction (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 3 (4) | 1 (1)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cerebral arteriovenous malformation haemorrhagic (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 3 (3)
Intestinal infarction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 3 (3) | 2 (2)
Death (General disorders) | 3 (3) | 4 (4)
Device dislocation (General disorders) | 1 (1) | 0 (0)
Device leakage (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 31 (31) | 17 (17)
Organ failure (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 3 (3) | 2 (2)
Sudden death (General disorders) | 3 (3) | 2 (2)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cytolytic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Candida sepsis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 2 (2)
Endocarditis pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis staphylococcal (Infections and infestations) | 2 (2) | 4 (4)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Fungal endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 6 (6)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 4 (4) | 8 (9)
Postoperative wound infection (Infections and infestations) | 2 (2) | 1 (1)
Prostatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyonephrosis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 2 (2)
Septic shock (Infections and infestations) | 7 (7) | 5 (5)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 18 (18) | 19 (19)
Staphylococcal infection (Infections and infestations) | 5 (5) | 5 (5)
Staphylococcal mediastinitis (Infections and infestations) | 8 (8) | 9 (9)
Staphylococcal osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 3 (3) | 2 (2)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 2 (2)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 4 (4) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Wound infection bacterial (Infections and infestations) | 2 (2) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 25 (25) | 27 (28)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraoperative cerebral artery occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Operative haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Cardiac output decreased (Investigations) | 1 (1) | 1 (1)
Troponin T increased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 3 (3)
Dizziness exertional (Nervous system disorders) | 0 (0) | 1 (1)
Encephalitis (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 2 (2)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 2 (2) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 3 (3)
Renal failure acute (Renal and urinary disorders) | 4 (4) | 2 (2)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (6)
Aneurysm ruptured (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Aortic rupture (Vascular disorders) | 1 (1) | 1 (1)
Aortic stenosis (Vascular disorders) | 2 (2) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis obliterans (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 3 (3) | 9 (9)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 3 (3) | 2 (2)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 4 (4)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V710 (60 µg) Lyophilized (N=3958) | Placebo (N=3967)
Injection site erythema (General disorders) | 280 (285) | 102 (104)
Injection site pain (General disorders) | 533 (575) | 232 (244)
Injection site swelling (General disorders) | 217 (222) | 79 (79)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.